CLINICAL TRIAL: NCT05574673
Title: Characterization of Epithelial Ovarian Cancer Patients in Terms of Homologous Recombination Phenotype - A Prospective Observational Study
Brief Title: Characterization of Epithelial Ovarian Cancer Patients in Terms of Homologous Recombination Phenotype
Acronym: HERO
Status: Recruiting | Type: Observational
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Other Study IDs: NSGO-CTU-HERO
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian cancer, observational study, HRD
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Kenny-Caffey syndrome, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer patients: Newly diagnosed patients with ovarian cancer, fallopian tube cancer or primary peritoneal cancer
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Patients receive standard of care treatment according to local and national guidelines

SUMMARY:
This is a prospective observational multi-country, multi-center study of a large real-world cohort of first line (1L) epithelial ovarian cancer patients, exposed to standard of care (SOC) treatment stratified according to BRCA1/2 and HRD status.

DETAILED DESCRIPTION:
The overall objective of the study is to demonstrate the distribution of ovarian cancer by HRD and BRCA1/2 mutational status and further characterize sub-cohorts of long- and short-term responders. Additionally, to collect representative clinical samples for further translational analyses.

The overall objective is separated by two distinct observational periods defined as Observational Period 1 (OP1) and Observational Period 2 (OP2):

* OP1: From date of diagnosis to date of first response assessment following 1L chemotherapy, progression or death, whichever occurs first
* OP2: From date of first response assessment following 1L chemotherapy to maximum 36 months following 1L chemotherapy, death or withdrawal of consent, whichever occurs first.

Objective for Observational Period 1 (OP1) The objective for OP1 is to demonstrate the distribution of ovarian cancer patients with FIGO stage I-II BRCA1/2mut ovarian cancer, or stage III-IV ovarian cancer in cohorts of BRCA1/2, HRD (either BRCA1/2 mutation and/or genomic instability), HRP and HR-unknown patients.

Objective for Observational Period 2 (OP2) The objective for OP2 is to further characterize sub-cohorts of short-term responders (progressing < 6 months following maintenance treatment) and long-term responders (progressing ≥ 32 months following maintenance treatment) in real-world cohorts of ovarian cancer patients. For FIGO stage I-II BRCA1/2mut or FIGO stage III-IV defined by HRD status determined by Myriad myChoice® CDx HRD test or non-Myriad local HRD test, and BRCA1/2 status.

A total of 350 patients will be enrolled from hospitals in Denmark, Finland, Norway, and Sweden. Competitive enrollment will be applied.

Eligible patients must have newly diagnosed histologically confirmed epithelial ovarian cancer:

* FIGO stage I-II with a known BRCA1/2 mutation (germline/gBRCA or somatic /tBRCA)
* FIGO stage III-IV of any histology of any histology.

ELIGIBILITY:
Patients are eligible to be included in the study, if all the following inclusion criteria are met:

* Patients with newly diagnosed histologically confirmed epithelial ovarian cancer:

  * FIGO stage I-II with a known BRCA1/2 mutation (germline/gBRCA or somatic/tBRCA)
  * FIGO stage III-IV of any histology
* Women aged ≥18 years of age at the time of diagnosis
* Patients intended for platinum-based chemotherapy treatment
* Patients capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Patients consent to provide archival tumor tissue sample

Patients are ineligible to be included in the study, if any of the exclusion criteria are met:

* Non-epithelial ovarian cancer, borderline tumors, or mucinous histology
* Patients with FIGO stage I-II, BRCAwt ovarian cancer

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed epithelial ovarian cancer patients (FIGO stage I-II with known BRCA1/2 mutation and FIGO stage III-IV of any histology), who are intended for 1L chemotherapy, will be recruited from specialist care centers across Denmark, Finland, Norway, and Sweden. In total 350 patients will be enrolled applying competitive enrollment. Each patient must meet all the inclusion criteria and none of the exclusion criteria to be included in the study. Under no circumstances can there be exceptions to this rule. Patients who do not meet the entry requirements are screen failures.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Endpoint OP1 | 36 months
  Frequency of surgical resection

SECONDARY OUTCOMES:
Endpoints OP1 - 1.1 | 36 months
  - First line anti-cancer treatment including outcome
Endpoints OP1 - 1.2 | 36 months
  - +/- Residual disease following Primary Cytoreductive Surgery (P-CRS)
Endpoints OP1 - 1.3 | 36 months
  - Overall Response Rate (ORR)
Endpoints OP1 - 1.4 | 36 months
  - BRCA1/2 and HRD status
Endpoint OP2 - 2.1 | 36 months
  - Number of patients receiving maintenance treatment or not
Endpoint OP2 - 2.2 | 36 months
  - Progression-Free-Survival (PFS) at 6, 12, 24 and 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Chair — NSGO-CTU
Locations (1):
- Rigshospitalet, København Ø, Region Sjælland, Denmark